CLINICAL TRIAL: NCT04632550
Title: Giant Left Atrium Atrial fibrillatioN CathEter Ablation, Posterior Box Isolation vs. Dallas Lesion Set: Prospective Randomized Trial (GLANCE Trial)
Brief Title: Giant Left Atrium Atrial fibrillatioN CathEter Ablation, Posterior Box Isolation vs. Dallas Lesion Set
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2020-0954
Record Dates: First submitted 2020-10-26; First posted 2020-11-17 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Population Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Circumferential pulmonary vein isolation(CPVI) group (Active Comparator)
  Interventions: Procedure: Circumferential pulmonary vein isolation(CPVI) group
- Posterior box isolation(POBI) group (Experimental)
  Interventions: Procedure: Posterior box isolation(POBI) group
- POBI+Anterior linear ablation(AL) group (Experimental)
  Interventions: Procedure: POBI+Anterior linear ablation(AL) group

INTERVENTIONS:
Procedure: Circumferential pulmonary vein isolation(CPVI) group — 1. PVI(pulmonary vein isolation) will be performed using a radiofrequency catheter
  2. Esophageal temperature will be monitored to prevent esophageal injury.
  3. Evaluation of procedure time, radiofrequency ablation time
  4. Evaluation of the complication after the procedure.
  5. Rhythm follow-up will be performed after the procedure in accordance with the aforementioned study design.
  Arms: Circumferential pulmonary vein isolation(CPVI) group
Procedure: Posterior box isolation(POBI) group — 1. PVI will be performed using a radiofrequency catheter
  2. Additional POBI(Posterior box isolation) is performed according to the traditional method and experience of the practitioner.
  3. Esophageal temperature will be monitored to prevent esophageal injury.
  4. The bidirectional block of each lesion set is the target of the procedures. But, we remain the incomplete block if three times of linear ablation failed to achieve the bidirectional block for the safety purpose.
  5. Evaluation of procedure time, radiofrequency ablation time
  6. Evaluation of the complication after the procedure.
  7. Rhythm follow-up will be performed after the procedure in accordance with the aforementioned study design.
  Arms: Posterior box isolation(POBI) group
Procedure: POBI+Anterior linear ablation(AL) group — 1. PVI, POBI will be performed using a radiofrequency catheter
  2. Additional AL(anterior linear) ablation is performed according to the traditional method and experience of the practitioner.
  3. Esophageal temperature will be monitored to prevent esophageal injury.
  4. The bidirectional block of each lesion set is the target of the procedures. But, we remain the incomplete block if three times of linear ablation failed to achieve the bidirectional block for the safety purpose.
  5. Evaluation of procedure time, radiofrequency ablation time
  6. Evaluation of the complication after the procedure.
  7. Rhythm follow-up will be performed after the procedure in accordance with the aforementioned study design.
  Arms: POBI+Anterior linear ablation(AL) group

SUMMARY:
Although the additional linear ablation after pulmonary vein isolation (PVI) is a class IIB indication for AF catheter ablation in patients with persistent AF, no clear benefit has been demonstrated in the recent randomized clinical trials (STAR-AF2 or POBI trials). Nevertheless, in the retrospective cohort data of this research team, additional POBI and AL were helpful in persistent AF patients with left atrial (LA) size > 50mm or more or low LA voltage. The purpose of this study was to evaluate the efficacy and safety of additional POBI and AL compared to CPVI alone in persistent AF patients with LA size over 50mm. Also, we intend to proceed with this randomized clinical trial with the high power short duration ablation protocol, which is effective in shortening the procedure time.

DETAILED DESCRIPTION:
A. Study design

1. Prospective randomization (pulmonary vein isolation [PVI] group vs. additional posterior box isolation [POBI] group vs. additional POBI and anterior line [AL] group)
2. Target number of subjects: 480 (160 per group)
3. Rhythm follow-up : 2012 ACC/AHA/ESC guidelines (Holter monitoring at the baseline, 2 month, and thereafter every 6 months; ECG if the patient has any symptom)
4. Anticoagulant therapy followed by 2014 ACC/AHA/ESC guidelines
5. All complications in each group will be evaluated including the re-hospitalization rate, major cardiovascular event, and mortality rate.

B. Progress and rhythm/ECG follow-up

1. To be performed in accordance with the 2012 ACC/AHA/HRS guidelines for AF management
2. Follow-up at 1 weeks, 3 months, and thereafter every 6-month after procedure.
3. Rhythm control at 3 months, and thereafter every 6-month follow-up with Holter
4. If the patient complains of symptoms, ECG will be performed at any time, and rhythm follow-up will be carried out with a Holter or event recorder.

C. Follow-up All the patients will be followed-up at 1, 3, 6 months, and thereafter every 6 months. If the patient shows any symptom within the clinical study period, patient will visit the outpatient clinic. ECG will be performed at every outpatient visits, and 24-hour Holter or event recording will be performed every 6 months for 2 years, and every year after 2 years (2012 Heart Rhythm Society/EHRA/European Cardiac Arrhythmia Society Expert Consensus Statement guidelines). If atrial fibrillation or atrial tachycardia lasting more than 30 seconds is observed in 12-lead ECG or Holter, it will be evaluated as recurrence. Recurrence within 3 months after the procedure will be classified as early recurrence, and that after 3 months will be classified as clinical recurrence.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with persistent atrial fibrillation who is scheduled for ablation procedure and ≥20 and ≤80 years of age
2. Left atrium size ≥ 50mm
3. Persistent atrial fibrillation that is recurrence during antiarrhythmic drug treatment or is not able to use an antiarrhythmic drug.
4. Patient who is indicated for anticoagulation therapy (for prevention of cerebral infarction)

Exclusion Criteria:

1. AF Patients with LA size less than 50mm
2. Atrial fibrillation associated with severe cardiac malformation or a structural heart disease that is hemodynamically affected
3. Patients with severe renal impairment or CT imaging difficulty using contrast media
4. Patients with a past history of radiofrequency ablation for atrial fibrillation or other cardiac surgery
5. Patients with active internal bleeding
6. Patients with contraindications for anticoagulation therapy(for prevention of cerebral infarction) and antiarrhythmic drugs
7. Patients with valvular atrial fibrillation (mitral stenosis >grade 2, mechanical valve, mitral valvuloplasty)
8. Patients with a severe comorbid disease
9. Expected survival < 1 year
10. Drug addicts or alcoholics
11. Patients who cannot read the consent form (illiterates, foreigners, etc.)
12. Other patients who are judged by the principal or sub-investigator to be ineligible for participation in this clinical study

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Safety evaluation: Procedure-related cardiac complication rate | within 30 days post procedure
  -including open cardiac surgery, cerebral infarction, pericardial effusion or cardiac tamponade, hematoma in the inguinal puncture site and vascular complications within 30 days post procedure.
Efficacy evaluation: clinical recurrence rate | Within 1 year after 3 months of procedure
  - Defined as atrial fibrillation or atrial tachycardia > 30 sec after 3 months within 1 year; based on the 2012 ACC/AHA/HRS guidelines, 24-hour Holter ECG monitoring will be performed at 2 month and every 6 months, and ECG and monitoring with a Holter or an event recorder will be performed at any time if the patient complains of symptoms
Efficacy evaluation: Major cardiovascular event rate | immediate after procedure
  - death, myocardial infarction, coronary angioplasty, and re-hospitalization for arrhythmia and heart failure
Efficacy evaluation: Major cardiovascular event rate | 12 months after procedure
  - death, myocardial infarction, coronary angioplasty, and re-hospitalization for arrhythmia and heart failure

SECONDARY OUTCOMES:
procedure time | immediate after the procedure
hospitalization duration | immediate after the discharge
Comparison of anti-arrhythmic drug or anticoagulation therapy related complication rate | immediate after the procedure, 1 week, 3,6,12,18,24,36 months after procedure.
rate of electrical cardioversion | immediate after the procedure, 1 week, 3,6,12,18,24,36 months after procedure.
rate of cardiovascular hospitalization | immediate after the procedure, 1 week, 3,6,12,18,24,36 months after procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Nam Pak, Principal Investigator — Severance Hospital
Locations (1):
- Yonsei Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided